CLINICAL TRIAL: NCT02655315
Title: Conservative Iron Chelation as a Disease-modifying Strategy in Parkinson's Disease. European Multicentre, Parallel-group, Placebo-controlled, Randomized Clinical Trial of Deferiprone"
Brief Title: Conservative Iron Chelation as a Disease-modifying Strategy in Parkinson's Disease
Acronym: FAIRPARKII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: European Commission (Other); ApoPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015_22; 2015-003679-31 (EudraCT Number); Grant agreement No 633190 (Other Grant/Funding Number: European Union's Horizon 2020); HP751 (Other: CTFG VHP)
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Deferiprone; Chelation
MeSH Terms: conditions — Parkinson Disease | interventions — Deferiprone; Bulk Drugs

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEFERIPRONE (Active Comparator): Half of participants will receive the deferiprone (DFP) to 15 mg / kg twice daily morning and evening (30mg / kg per day).The treatment lasts nine months.
  Interventions: Drug: Deferiprone
- PLACEBO (Placebo Comparator): Half of participants will receive the placebo twice daily morning and evening. The treatment lasts nine months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deferiprone — 15 mg / kg twice daily morning and evening (30mg / kg per day).The treatment lasts nine months.
  Other Names: active drug
  Arms: DEFERIPRONE
Drug: Placebo — the placebo twice daily morning and evening. The treatment lasts nine months
  Other Names: harmless pill; inactive drug
  Arms: PLACEBO

SUMMARY:
This study evaluates the effect of iron chelation as a therapeutic strategy to slow the progression of Parkinson's disease. Half of participants will receive the deferiprone to 15 mg / kg twice daily morning and evening (30mg / kg per day), while the other half will receive a placebo. The treatment lasts nine months.

DETAILED DESCRIPTION:
This is the new concept of "conservative iron chelation". We recently demonstrated (for the first time) the feasibility, efficacy and acceptability of the conservative iron chelation approach in pilot translational studies in Parkinson's disease with a prototype drug: deferiprone (1,2-dimethyl-3-hydroxypyridin-4-one) (in the FAIR-PARK-I project led by the applicant and funded by French Ministry of Health). The only available blood-brain-barrier-permeable iron chelator deferiprone is approved for treating systemic iron overload in transfused patients with thalassemia. Deferiprone has been on the European Union market since 1999, with a favourable risk/benefit balance at dose of 75 to 100 mg/kg/day. The investigators shall adopt a repositioning strategy by using deferiprone at a lower dose of 30 mg/kg/day in this new indication for local iron overload in Parkinson's disease. Deferiprone will be the first-in-class drug for this novel therapeutic strategy. On the basis of the preclinical and clinical data from (FAIR-PARK-I), the present (FAIR-PARK-II) project should constitute a model for future cytoprotection strategies in neurodegenerative diseases; if deferiprone treatment is associated with significant slower disease progression, it would be the first non-dopaminergic drug to have a proven disease-modifying effect in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Parkinson's disease diagnosed according United Kingdom Parkinson's disease Society Brain Bank Clinical Diagnostic Criteria and based on the presence of at least two of the three cardinal features of the disease (rest tremor, bradykinesia and rigidity). If rest tremor is not present, subjects must have unilateral onset of symptoms.
3. Treatment-naïve, i.e. the best population for assessing a disease-modifying effect without the interaction of dopaminergic treatment (no dopaminergic agonists, L-dopa, anticholinergics, monoamine oxidase B inhibitors (e.g. rasagiline) or deep brain stimulation).
4. Patients covered by a Health Insurance System in countries where required by law
5. Written informed consent dated and signed prior to the beginning of any procedures related to the clinical trial

Exclusion Criteria:

1. Disease duration greater than 18 months.
2. Patients with high frequency of comorbidity or vital risks that may reasonably impair life expectancy
3. Subject with handicap required dopaminergic treatment at the inclusion and therefore likely not to bear 9 months without symptomatic treatment
4. Hoehn and Yahr stage 3 or more.
5. Significant cognitive impairment (a Mini Mental State Examination score <24 or an equivalent impairment on a similar scale) or dementia diagnosed in accordance with the Movement Disorders Society criteria (Emre et al., 2007).
6. Atypical or secondary parkinsonism (supranuclear palsy, multisystem atrophy, etc.) or anomalies on MRI suggestive of vascular involvement or significant cortical or subcortical atrophy (i.e. atypical for Parkinson's Disease).
7. Progressing axis I psychiatric disorders (psychosis, hallucinations, substance addiction, bipolar disorder, or severe depression), in accordance with the Diagnostic and Statistical Manual of Mental Disorders.
8. Subjects undergoing brain stimulation.
9. Positive Human Immunodepression Virus serology.
10. Hypersensitivity to deferiprone.
11. Patients with agranulocytosis or with a history of agranulocytosis.
12. Patients taking a treatment at risk of agranulocytosis (clozapine, Closaril®/Leponex®).
13. Patients with anaemia (regardless of the latter's aetiology) or a history of another haematological disease. Haemochromatosis is not an exclusion criterion.
14. Pregnant or breastfeeding women or women of childbearing potential not taking highly effective contraception.
15. Kidney or liver failure.
16. Other serious diseases.
17. Inability to provide informed consent.
18. Participation in another clinical trial with investigational medicinal product within 3 months prior to inclusion in the study
19. Patient who has suffered mild or moderate depressive episode and isn't in remission and on a stable medication for at least 8 weeks
20. Patient > 130k

Exclusion criteria for the biomarker study and the ancillary study (i) Magnetic Resonance Imaging:

* Subjects for whom Magnetic Resonance Imaging is contraindicated (metal objects in the body, severe claustrophobia, pacemaker, incompatible surgical material).
* Very severe rest tremor, which could induce Magnetic Resonance Imaging artefacts.

(ii) Lumbar puncture:

* Blood coagulation disorders, antiplatelet drugs or anticoagulants.
* Intracranial hypertension. (iii) Contraindications to nitrous oxide:
* Ventilation with Fraction of inspired Oxygen >50%, emphysema or pneumothorax
* Altered states of consciousness, non-cooperative patient (need to stop the nitrous oxide)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Global effect (symptomatic and disease modifying effects) on motor and non motor handicap | at 36 weeks
  the change in the total Movement Disorders Society-Unified Parkinson Disease Rating Scale score between baseline and 36 weeks (i.e. the end of the placebo-controlled phase for analysis of both disease-modifying and symptomatic effects)

SECONDARY OUTCOMES:
Disease-modifying effect on motor and non motor handicap | baseline, at 40 weeks
  It will be measured as the changes in the overall Movement Disorders Society-Unified Parkinson Disease Rating Scale score between baseline and week 40 (i.e. the end of the one-month post-treatment monitoring period), to analyse the disease-modifying effect without bias from the symptomatic effect of ongoing deferiprone treatment) on the study population
Effect of the motor symptoms | baseline, at 12, 36 and 40 weeks
  The effect of the motor symptoms will be analysed as the change in the subscale part III of the Movement Disorders Society-Unified Parkinson Disease Rating Scale score
Quality of life and autonomy by PDQ-39 score | baseline, at 36 and 40 weeks
  It will be analyzed as the change in the Parkinson's Disease Quality of Life (PDQ-39, via a 39-item self-questionnaire)
Quality of life and autonomy by Clinical Global Impression score | baseline, at 36 and 40 weeks
  the Clinical Global Impression scored by the examiner and the patient
Health economics assessment | baseline, at 36 and 40 weeks
  will be performed via a specific questionnaire provides a simple descriptive profile and a single index value for health status
EQ-5D questionnaire | baseline, at 36 and 40 weeks
  the questionnaire provides a simple descriptive profile and a single index value for health status.
Safety criteria | 40 weeks
  All the safety concerns will be listed in a table with the number of patients, the type the severity and the time of occurrence for
  * adverse events
  * neutropenia (weekly complete blood count)
  * agranulocytosis (weekly complete blood count)
  * anemia (weekly complete blood count)
  * iron metabolism abnormalities (haemoglobin, serum iron, ferritinemia, transferrin, total binding capacity, transferrin saturation coefficient, 24-hour urine iron).
  * Standard biological abnormalities (fasting glucose, urea, creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and (for all sexually active, fertile females) urine pregnancy tests.
  * Abnormal physical examination (including vital signs, bodyweight, electrocardiogram and blood pressure)
Effect on overall cognitive status | baseline, at 12, 36 and 40 weeks
  Measured by the score in the Montreal Cognitive Assessment
Effect on gait disorders | baseline, at 12, 36 and 40 weeks
  Measured by the Stand Walk Sit test
Effect on daily living | baseline, at 12, 36 and 40 weeks
  The effect on daily living will be analysed as the change in the subscale part II (activities of daily living) of the Movement Disorders Society-Unified Parkinson Disease Rating Scale score
Effect on non-motor symptoms | baseline, at 12, 36 and 40 weeks
  The effect on non motor symptoms will be analysed as the change in the subscale part I (cognition and behavior) of the Movement Disorders Society-Unified Parkinson Disease Rating Scale score
Lack of occurrence of motor fluctuations | baseline, at 12, 36 and 40 weeks
  The lack of occurrence of motor fluctuations will be analysed on the subscale part IV of the Movement Disorders Society-Unified Parkinson Disease Rating Scale score

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Study Chair — University Hospital, Lille
Locations (25):
- Medizinische Universitat Innsbruck, Innsbruck, Austria
- Czechia (2):
  - Charles University, Prague
  - Univerzita Karlova V Praze, Prague
- France (8):
  - CHU Pellegrin, Bordeaux
  - Hôpital Wertheimer, Bron
  - Hôpital Montpied, Clermont-Ferrand
  - Hôpital Salengro, CHRU, Lille
  - CHU la TIMONE, Marseille
  - AP-HP, Hôpital Pitié-Salpêtrière, Paris
  - CHU de Strasbourg, Hôpital de Hautepierre, Strasbourg
  - Chu Purpan, Toulouse
- Germany (3):
  - University Hospital, Saarland University, Homburg
  - Christian-albrechts universität zu kiel, Kiel
  - Klinik und Poliklinik für Neurologie der Universitätsmedizin Rostock, Rostock
- Netherlands (2):
  - Acadamic central center, Amsterdam, Amsterdam
  - Radboud university medical center, Nijmegen
- Portugal (3):
  - Centro Hospitalar e universitario de Coimbra, Coimbra
  - Centro Hospitalar do Alto Ave, Guimarães
  - Centro Hospitalar Lisboa Norte, Lisbon
- Spain (3):
  - Hospital Clinic Universitari de Barcelona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
- United Kingdom (3):
  - Cambridge University Hospital, Cambridge
  - University of Glasgow, Glasgow
  - Newcastle University, Newcastle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Devos D, Labreuche J, Rascol O, Corvol JC, Duhamel A, Guyon Delannoy P, Poewe W, Compta Y, Pavese N, Ruzicka E, Dusek P, Post B, Bloem BR, Berg D, Maetzler W, Otto M, Habert MO, Lehericy S, Ferreira J, Dodel R, Tranchant C, Eusebio A, Thobois S, Marques AR, Meissner WG, Ory-Magne F, Walter U, de Bie RMA, Gago M, Vilas D, Kulisevsky J, Januario C, Coelho MVS, Behnke S, Worth P, Seppi K, Ouk T, Potey C, Leclercq C, Viard R, Kuchcinski G, Lopes R, Pruvo JP, Pigny P, Garcon G, Simonin O, Carpentier J, Rolland AS, Nyholm D, Scherfler C, Mangin JF, Chupin M, Bordet R, Dexter DT, Fradette C, Spino M, Tricta F, Ayton S, Bush AI, Devedjian JC, Duce JA, Cabantchik I, Defebvre L, Deplanque D, Moreau C; FAIRPARK-II Study Group. Trial of Deferiprone in Parkinson's Disease. N Engl J Med. 2022 Dec 1;387(22):2045-2055. doi: 10.1056/NEJMoa2209254. PMID 36449420
- [Derived] Mahoney-Sanchez L, Bouchaoui H, Ayton S, Devos D, Duce JA, Devedjian JC. Ferroptosis and its potential role in the physiopathology of Parkinson's Disease. Prog Neurobiol. 2021 Jan;196:101890. doi: 10.1016/j.pneurobio.2020.101890. Epub 2020 Jul 26. PMID 32726602
- [Derived] Moreau C, Duce JA, Rascol O, Devedjian JC, Berg D, Dexter D, Cabantchik ZI, Bush AI, Devos D; FAIRPARK-II study group. Iron as a therapeutic target for Parkinson's disease. Mov Disord. 2018 Apr;33(4):568-574. doi: 10.1002/mds.27275. Epub 2018 Jan 30. No abstract available. PMID 29380903
- See also: Website for informations on the Fairpark2 study — http://fairpark2.eu/